CLINICAL TRIAL: NCT02751229
Title: Adaptation and Evaluation of the Honest Open Proud Program for Adolescents With Mental Illness
Brief Title: Honest Open Proud for Adolescents With Mental Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Child and Adolescent Psychiatry Weissenau, Centre for Psychiatry in South-Württemberg, Germany (Unknown); Josefinum, Child and Adolescent Psychiatry and Psychotherapy, Augsburg, Germany (Unknown); Illinois Institute of Technology, Chicago, USA (Unknown)
Responsible Party: Principal Investigator, Nicolas Rüsch, Professor, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOP-Adolescents
Record Dates: First submitted 2016-03-24; First posted 2016-04-26 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Secrecy Versus Disclosure Among Adolescents With Mental Illness
Keywords: Mental illness; adolescents; intervention; stigma; disclosure; secrecy
MeSH Terms: conditions — Mental Disorders; Social Stigma

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Honest Open Proud (Experimental): The group program is about disclosure ('coming out') versus secrecy of one's mental illness. The groups are facilitated by peers (young adults with mental illness) and mental health professionals. Each group runs for three weeks, one meeting per week, and two hours per meeting.
  Fidelity to manual: rated by PhD student in each session as proportion of key topics covered
  Interventions: Behavioral: Honest Open Proud (HOP)
- Control Group (No Intervention): treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Honest Open Proud (HOP) — five lessons in three modules, two for each two-hour session
  1. Considering pros and cons of disclosing:
     * hurtful and helpful attitudes about mental illness
     * identify beliefs participants hold about themselves
     * explore five-step process to challenge their personally hurtful beliefs
     * weigh pros and cons of coming out in order to facilitate a decision on whether to disclose
  2. Different ways to disclose:
     * different levels of (non-) disclosure and how to weigh the cons and pros
     * disclosure via social media versus disclosing face to face
     * how to find people that are better to disclose to than others and how to 'test them out'
     * participants will discuss how others might respond to their disclosure and how that will affect them
  3. Telling your story:
     * how to tell one's story in a personally meaningful way, how to identify peers who might help with the coming out process, to review how telling one's story felt
  Other Names: Coming Out Proud (COP)
  Arms: Honest Open Proud

SUMMARY:
The purpose of the study is to evaluate the efficacy of the group-based intervention 'Honest Open Proud' among adolescents with mental illness.

DETAILED DESCRIPTION:
Both due to fear of public stigma and due to self-stigma or shame, people with mental illness may decide to keep their condition a secret or even to withdraw from other people altogether in order to minimise the risk of being labelled. Secrecy can help on the short term to protect individuals from public stigma, but often it has negative long-term consequences such as social isolation, distress and unemployment. Disclosure, on the other hand, carries the risk to be discriminated by others, but can reduce the burden of secrecy, lead to support by others and reduce public stigma. In this study investigators aim to evaluate whether a group program run both by people with mental illness (peers) and professionals helps to reduce self-stigma and makes it easier for adolescents to handle the necessary choices related to secrecy versus disclosure.

ELIGIBILITY:
Inclusion Criteria:

* At least one self-reported current axis I or axis II disorder according to DSM-5 (American Psychiatric Association, 2013), which is not restricted to only substance-related disorder(s)
* Age 13 to 18
* Ability to provide written informed consent
* Fluid in German (needed for self-report measures)
* At least a moderate level of self-reported disclosure-related distress/difficulty (score 4 or higher on the screening item 'In general, how distressed or worried are you in terms of secrecy or disclosure of your mental illness to others?', rated from 1, not at all, to 7, very much)

Exclusion Criteria:

* Self-reported diagnosis of only a substance- or alcohol-related disorder, without non-substance related current psychiatric comorbidity. We will exclude people who only have a substance-/alcohol-related disorder because the disclosure of these disorders is not the topic of the HOP intervention
* Intellectual disability
* Organic disorders

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Stigma Stress Scale, 8 items (Rüsch, Corrigan, Wassel et al., 2009; Rüsch, Corrigan, Powell et al., 2009) | 3 weeks (T1)
Health-Related Quality of Life Questionnaire KIDSCREEN-10 Index, 10 items (Deighton et al., 2014; Ravens-Sieberer et al., 2010) | 6 weeks (T2)

SECONDARY OUTCOMES:
Satisfaction with intervention questionnaire (according to Keller, Konopka, Fegert, & Naumann, 2003; own development) | 3 weeks
Empowerment Scale, Subscales 'self-esteem' and 'control over the future', 13 items (Rogers, Chamberlin, Ellison, & Crean, 1997) | baseline, 3 and 6 weeks
Attitudes to disclosure, 2 items (Rüsch, Evans-Lacko, Henderson, Flach, & Thornicroft, 2011) | baseline, 3 and 6 weeks
  2 items on attitudes to disclosure, adapted from a UK Dept of Health survey (see above Rüsch et al 2011 reference for further details) with seven-point Likert scale
Disclosure Distress, 1 item ("In general, how distressed or worried are you in terms of secrecy or disclosure of your mental illness to others?', from 1, not at all, to 7, very much) (Rüsch et al., 2014a) | baseline, 3 and 6 weeks
Shame about having a mental illness, 1 item ("Do you feel ashamed about having a mental illness?"; from 1, not at all, to 7, very much) (Rüsch et al., 2014b) | baseline, 3 and 6 weeks
General Help-Seeking Questionnaire, 1 item (Wilson et al., 2005) | baseline, 3 and 6 weeks
Beck Hopelessness Scale (BHS), 4-item short version (Yip, Paul S F & Cheung, 2006) | baseline, 3 and 6 weeks
Self-Stigma of Mental Illness Scale (SSMIS), Subscale 'self-concurrence', 5 items (Corrigan et al., 2012; Rüsch et al., 2006) | baseline, 3 and 6 weeks
Self-Identified Stage of Recovery (SISR), 5 items (Andresen, Caputi, & Oades, 2010) | baseline, 3 and 6 weeks
  brief self-rated assessment of stage of recovery; consists of two parts (A & B): Part A reflects five statements about stages of recovery, participants have to choose one that best reflects their current experience. Part B consists of four statements reflecting recovery processes, rated on a six-point Likert scale
Internalised Stigma of Mental Illness Inventory (ISMI), 10-item short version (Boyd, Otilingam, & Deforge, 2014) | baseline, 3 and 6 weeks
Social withdrawal and secrecy, 12 item-short version (Link et al., 2009) | baseline, 3 and 6 weeks

OTHER OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D), 15 items (Meyer & Hautzinger, 2001) | baseline, 3 and 6 weeks
Strengths and Difficulties Questionnaire (SDQ), Subscale 'peer relationship problems', 5 items (Goodman, 2001) | baseline, 3 and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rüsch, Professor, Principal Investigator — Department of Psychiatry II, Section Public Mental Health, Ulm University, Bezirkskrankenhaus Günzburg, Germany
Locations (5):
- Illinois Institute of Technology, Chicago, Illinois, United States
- Germany (4):
  - Josefinum, Child and Adolescent Psychiatry and Psychotherapy, Augsburg
  - Department of Psychiatry II, Section Public Mental Health, Ulm University, Bezirkskrankenhaus Günzburg, Ulm
  - Child and Adolescent Psychiatry and Psychotherapy, University of Ulm, Ulm
  - Child and Adolescent Psychiatry Weissenau, Centre for Psychiatry in South-Württemberg, Weißenau

REFERENCES:
- [Background] Andresen R, Caputi P, Oades LG. Do clinical outcome measures assess consumer-defined recovery? Psychiatry Res. 2010 May 30;177(3):309-17. doi: 10.1016/j.psychres.2010.02.013. Epub 2010 Mar 15. PMID 20227768
- [Background] Boyd JE, Otilingam PG, Deforge BR. Brief version of the Internalized Stigma of Mental Illness (ISMI) scale: psychometric properties and relationship to depression, self esteem, recovery orientation, empowerment, and perceived devaluation and discrimination. Psychiatr Rehabil J. 2014 Mar;37(1):17-23. doi: 10.1037/prj0000035. PMID 24660946
- [Background] Corrigan PW, Michaels PJ, Vega E, Gause M, Watson AC, Rusch N. Self-stigma of mental illness scale--short form: reliability and validity. Psychiatry Res. 2012 Aug 30;199(1):65-9. doi: 10.1016/j.psychres.2012.04.009. Epub 2012 May 10. PMID 22578819
- [Background] Deighton J, Croudace T, Fonagy P, Brown J, Patalay P, Wolpert M. Measuring mental health and wellbeing outcomes for children and adolescents to inform practice and policy: a review of child self-report measures. Child Adolesc Psychiatry Ment Health. 2014 Apr 29;8:14. doi: 10.1186/1753-2000-8-14. eCollection 2014. PMID 24834111
- [Background] Ravens-Sieberer U, Erhart M, Rajmil L, Herdman M, Auquier P, Bruil J, Power M, Duer W, Abel T, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J; European KIDSCREEN Group. Reliability, construct and criterion validity of the KIDSCREEN-10 score: a short measure for children and adolescents' well-being and health-related quality of life. Qual Life Res. 2010 Dec;19(10):1487-500. doi: 10.1007/s11136-010-9706-5. Epub 2010 Jul 30. PMID 20668950
- [Background] Rogers ES, Chamberlin J, Ellison ML, Crean T. A consumer-constructed scale to measure empowerment among users of mental health services. Psychiatr Serv. 1997 Aug;48(8):1042-7. doi: 10.1176/ps.48.8.1042. PMID 9255837
- [Background] Rusch N, Corrigan PW, Heekeren K, Theodoridou A, Dvorsky D, Metzler S, Muller M, Walitza S, Rossler W. Well-being among persons at risk of psychosis: the role of self-labeling, shame, and stigma stress. Psychiatr Serv. 2014 Apr 1;65(4):483-9. doi: 10.1176/appi.ps.201300169. PMID 24382666
- [Background] Rusch N, Corrigan PW, Powell K, Rajah A, Olschewski M, Wilkniss S, Batia K. A stress-coping model of mental illness stigma: II. Emotional stress responses, coping behavior and outcome. Schizophr Res. 2009 May;110(1-3):65-71. doi: 10.1016/j.schres.2009.01.005. Epub 2009 Feb 23. PMID 19237266
- [Background] Rusch N, Corrigan PW, Wassel A, Michaels P, Olschewski M, Wilkniss S, Batia K. A stress-coping model of mental illness stigma: I. Predictors of cognitive stress appraisal. Schizophr Res. 2009 May;110(1-3):59-64. doi: 10.1016/j.schres.2009.01.006. Epub 2009 Mar 6. PMID 19269140
- [Background] Rusch N, Evans-Lacko SE, Henderson C, Flach C, Thornicroft G. Knowledge and attitudes as predictors of intentions to seek help for and disclose a mental illness. Psychiatr Serv. 2011 Jun;62(6):675-8. doi: 10.1176/ps.62.6.pss6206_0675. PMID 21632739
- [Background] Rusch N, Holzer A, Hermann C, Schramm E, Jacob GA, Bohus M, Lieb K, Corrigan PW. Self-stigma in women with borderline personality disorder and women with social phobia. J Nerv Ment Dis. 2006 Oct;194(10):766-73. doi: 10.1097/01.nmd.0000239898.48701.dc. PMID 17041289
- [Background] Wilson, CJ, Deane, FP, Ciarrochi, J, Rickwood, D. Measuring help-seeking intentions: Properties of General Help-Seeking Questionnaire. Canadian Journal of Counselling, 39(1), 15-28, 2005.
- [Background] Yip PS, Cheung YB. Quick assessment of hopelessness: a cross-sectional study. Health Qual Life Outcomes. 2006 Mar 1;4:13. doi: 10.1186/1477-7525-4-13. PMID 16509984
- [Background] Keller, F, Konopka, L, Fegert, JM, Naumann, A . Prozessaspekte der Zufriedenheit von Jugendlichen in stationär-psychiatrischer Behandlung [Patient satisfaction of adolescents during in-patient psychiatric treatment: a process-oriented approach]. Nervenheilkunde 22: 40-46, 2003.
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Meyer, TD, & Hautzinger, M. Allgemeine Depressions-Skala (ADS) [Center for Epidemiological Studies - Depression Scale (CES-D) - Norms for adolescents and extension for the assessment of manic symptoms]. Diagnostica, 47(4): 208-215, 2001.
- [Background] Rusch N, Abbruzzese E, Hagedorn E, Hartenhauer D, Kaufmann I, Curschellas J, Ventling S, Zuaboni G, Bridler R, Olschewski M, Kawohl W, Rossler W, Kleim B, Corrigan PW. Efficacy of Coming Out Proud to reduce stigma's impact among people with mental illness: pilot randomised controlled trial. Br J Psychiatry. 2014;204(5):391-7. doi: 10.1192/bjp.bp.113.135772. Epub 2014 Jan 16. PMID 24434073
- [Derived] Mulfinger N, Muller S, Boge I, Sakar V, Corrigan PW, Evans-Lacko S, Nehf L, Djamali J, Samarelli A, Kempter M, Ruckes C, Libal G, Oexle N, Noterdaeme M, Rusch N. Honest, Open, Proud for adolescents with mental illness: pilot randomized controlled trial. J Child Psychol Psychiatry. 2018 Jun;59(6):684-691. doi: 10.1111/jcpp.12853. Epub 2017 Dec 5. PMID 29205343